CLINICAL TRIAL: NCT06776640
Title: Efficacy of Perioperative Oral Vitamin D3 Supplementation on Implant Osseointegration in Patients With Vitamin D Deficiency
Brief Title: Perioperative Oral Vitamin D3 Supplementation on Implant Osseointegration
Acronym: OSIVID
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_AGC_osivid_001
Record Dates: First submitted 2024-12-20; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Implant Site Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with supplementation of vitamin D3: perioperative oral vitamin D3 supplementation on implant osseointegration in patients with vitamin D deficiency.

SUMMARY:
The number of patients treated in Implantology at Nantes University Hospital is 400 per year. This pilot study aims to demonstrate the efficacy of a 6-month oral cholecalciferol supplementation on osseointegration in patients requiring dental implants and presenting with vitamin D deficiency, compared to French patients who have not undergone vitamin D screening

DETAILED DESCRIPTION:
This study will be conducted on patients with vitamin D deficiency or insufficiency who visit the Restorative and Surgical Dentistry Department at the Dental Care Center of Nantes University Hospital for implant surgery. The investigator will present the study to them and record their verbal non-opposition. Clinical data from before the surgery (approximately 3 months prior), during the surgery, and postoperative visits up to 3 months afterward will be included in the OSIVID study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥ 18 years old, candidate for dental implant placement.
* with vitamin D deficiency or insufficiency: 25(OH)D < 25 ng/L.
* affiliated with a social security scheme.

Exclusion Criteria:

* with a local contraindication for implant placement.
* under guardianship, curatorship, or legal protection
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted on patients with vitamin D deficiency or insufficiency who visit the Restorative and Surgical Dentistry Department at the Dental Care Center of Nantes University Hospital for implant surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
The stability of the implan | 3 months (surgery and 3 months after)
  The stability of the implant measured by RFA (Resonance Frequency Analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Gaelle Chaux, MD PhD, Principal Investigator — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: Undecided